CLINICAL TRIAL: NCT00753246
Title: Phase-III Study of Standard Radiotherapy Plus Concomitant and Adjuvant OSAG 101 (Theraloc®) Plus Temozolomide vs. Standard Radiotherapy Plus Concomitant and Adjuvant Temozolomide in Patient With Newly Diagnosed, Histologically Confirmed Glioblastoma Multiforme Grade IV
Brief Title: Nimotuzumab in Adults With Glioblastoma Multiforma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oncoscience AG (Industry)
Collaborators: Neurological Clinic, Knappschaftskrankenhaus Bochum-Langendreer, Bochum, Germany (Unknown); University of Bonn (Other); Dep. of Neurosurgery and Policlinic, University Hospital, Dresden, Germany (Other); Heinrich-Heine University, Duesseldorf (Other); Johann Wolfgang Goethe University Hospital (Other); University of Giessen (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Kiel (Other); Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other); Universität Tübingen (Other)
Responsible Party: Oncoscience AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSAG101-BSA05
Record Dates: First submitted 2007-11-20; First posted 2008-09-16 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Adults With Glioblastoma Multiforma
Keywords: glioblastoma multiforma
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Placebo Comparator): adults with TMZ, RT
  Interventions: Drug: nimotuzumab
- Arm A (Experimental): adults with TMZ, RT, nimotuzumab
  Interventions: Drug: nimotuzumab

INTERVENTIONS:
Drug: nimotuzumab — monoclonal antibody

SUMMARY:
Determination of efficiency of nimotuzumab in adults with glioblastoma multiforma

DETAILED DESCRIPTION:
The objective of the present study is a comparison of treatment of patients with newly diagnosed glioblastoma multiforme grade IV. Patients will be randomized in one of two arms when included. Patients randomly assigned to arm A will receive Nimotuzumab (OSAG 101) plus Temozolomide concomitant with standard radiotherapy. Patients randomised in arm B will receive standard radiotherapy plus Temozolomide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent
* Newly diagnosed, histologically confirmed glioblastoma multiforme grade IV
* Condition is measurable by MRI in at least one dimension
* Age 18-70
* Karnofsky-Index > 40
* Treatment in a study center
* Female patients with a childbearing potential must have a negative pregnancy test within one week before inclusion in the trial. Those female and male patients admitted in the study must use a reliable method of contraception.
* Adequate haematological, renal and hepatic function:

  * Leucocytes >2.0x10^9/l
  * Hb> 10g/dl
  * Billirubin total < 2.5x upper limit of normal (ULN)
  * Creatinin i.S. < 1.5x ULN
  * AST (GOT)/ALT (GPT) < 5x ULN

Exclusion Criteria:

* Patients with history of anaphylactic reaction to murine or humanized antibody
* Patients with evidence second malignancy
* Patients who are pregnant or patients who refused adequate contraceptive precaution (female and male) during the trial
* Pregnancy and lactation
* Other conditions considered by investigators as sound reasons for disqualification from enrolment into the study such as: potential non compliance with protocol requirement
* No MRI for tumour evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-08; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Progression-free interval determined by MRI | week 12, 24, 36, 52

SECONDARY OUTCOMES:
Overall survival Time to reintervention Response rate according to RECIST criteria Toxicity according to CTC criteria Symptom control Quality of life | week 12, 24, 36, 52

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Westphal, Prof. MD, Principal Investigator — University Hamburg
Locations (1):
- Dep. Neurosurgery, Univ. Hamburg, Hamburg, Germany